CLINICAL TRIAL: NCT05794451
Title: Developing an Artificial Intelligence System to Detect Mild Cognitive Impairment and Alzheimer's Disease Dementia Through Self-Figure Drawing: An Innovative Approach
Brief Title: Developing an Artificial Intelligence System to Detect Cognitive Impairment
Status: Recruiting | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Johanna Czamanski-Cohen, Senior Lecturer, University of Haifa
Other Study IDs: ALZAI
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Healthy Aging; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: Adults aged 60 and above without cognitive impairment
- Mild cognitive impairment: Adults 60 and above with mild cognitive impairment
- Alzheimer's disease: Adults diagnosed with Alzheimer's disease

SUMMARY:
Alzheimer's disease dementia (AD) is a debilitating and prevalent neurodegenerative disease in older adults globally. Cognitive impairment, a hallmark of AD, is assessed through verbal tests that require high specialization, and while accepted as screening tools for AD, general practitioners seldom use them. AD can be diagnosed with expensive, invasive neuroimaging and blood tests, but these are usually conducted when cognitive functioning is already severely impaired. Thus, finding a novel, non-invasive tool to detect and differentiate mild cognitive impairment (MCI) and AD is a prime public health interest. Self-figure drawings (a projective tool in which individuals are asked to draw a picture of themselves), are easy to administer and have been shown to differentiate between healthy and cognitively impaired individuals, including AD. Convolutional Neural Network (CNN) (a type of deep neural network, applied to analyze visual imagery) has advanced to assess health conditions using art products. Therefore, the proposed study suggests utilizing CNN-based methods to develop and test an application tailored to differentiate between drawings of individuals with MCI, AD, and healthy controls (HC) using 4,000 self-figure drawings. This

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 and above with subtle signs of risk of future cognitive decline, residing in the community or in nursing homes with a minimum of 10 years of education.

Exclusion Criteria:

* Current or past psychiatric illness, the presence of congenital/organic cognitive condition, severe visual or motor impairment, and terminal illness (to avoid the effect of comorbidities).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 60 or above, who live in Israel.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognition | One day
  The Montreal Cognitive Assessment (MoCA) is a 10-minute paper-based test that aims to detect MCI in older patients with symptomatology, suggesting impaired cognition. The MoCA is composed of 12 tasks to detect short-term memory, visuospatial ability, executive functioning, phonemic fluency, abstraction, attention, concentration, working memory, language, and orientation.
Cognition for adults diagnosed with Alzheimer's disease | One day
  The Self-reported Cognitive Difficulties (CDS)75 is a 39-item questionnaire that requires participants or their caregivers in case of AD to rate how often they currently experience cognitive difficulties in everyday life using a 5-point scale (0 -"never" to 4 -"very often").
Self-figure drawing -Cognition | One day
  Self-figure drawing. Participants will be asked to draw themselves using a pencil on an A4-sized sheet of paper.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Czamanski-Cohen, PhD, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
This is an artificial intelligence study, thus there will not be a dataset available for sharing.